CLINICAL TRIAL: NCT05438472
Title: Incidence, Patient Characteristics and Outcome of Myocarditis After COVID-19 mRNA Vaccine (MACIS)
Brief Title: Incidence, Patient Characteristics and Outcome of Myocarditis After COVID-19 mRNA Vaccine
Acronym: MACIS
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-02339; kt22Mueller
Record Dates: First submitted 2022-06-29; First posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Myocarditis
Keywords: Major Adverse Cardiac Events (MACE); COVID-19 vaccination; Comirnaty (Pfizer/BioNTech) mRNA vaccine; Moderna mRNA vaccine; myopericarditis; health care professionals; COVID-19 booster vaccination; vaccination-induced myocarditis
MeSH Terms: conditions — Myocarditis; Cardiovascular Diseases | interventions — Data Collection; Health Personnel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- healthcare professionals with COVID-19 mRNA vaccine booster: Consecutive individuals that received a COVID-19 mRNA vaccine booster and undergo a systematic approach to detect myocarditis at the University Hospital Basel. The project population includes mainly healthcare workers, aged between 16-65, most of them with presumable no comorbidities. Baseline characteristics include age, divided in several groups (16-20 years, 21-25 years, 26-30 years, 31-35 years, 36-40 years, 41-45 years, 46-50 years, 51-55 years, 56-60 years, 61-65 years).
  Interventions: Other: data collection in healthcare professionals with COVID-19 mRNA vaccine booster

INTERVENTIONS:
Other: data collection in healthcare professionals with COVID-19 mRNA vaccine booster — Day 3 (48 - 96h) post COVID-19 mRNA booster: data collection on symptoms (chest pain, dyspnea, myalgia, fever, chills); blood sample for cardiomyocyte injury (hs-cTnT, hs-cTnI). If elevated hs-cTnT concentration, participant has to avoid strenuous exercise. Work-up on Day 4: clinical evaluation, ECG, 2. blood sampling for hs-cTnT. If hs-cTnT > 100 ng/l, cardiac magnetic resonance imaging is done for signs of cardiac inflammation. If hs-cTnT rises above upper limit but doesn't exceed 100 ng/l, clinical exam might be evaluated. In confirmed myocarditis, a clinical assessment (treatment, need for hospitalization, length of rhythm monitoring, rest) is evaluated by a cardiologist. Day 4: EDTA blood from all subjects with elevated troponin at day 3 post-vaccination is collected for pathomechanism of mRNA vaccine associated myocarditis. 1-month follow-up: questionnaire on predefined cardiac endpoints.

SUMMARY:
This study evaluates the incidence, patient characteristics and outcome of myocarditis after the COVID-19 mRNA vaccination in healthcare professionals.

DETAILED DESCRIPTION:
Considering previous reports of cardiovascular adverse events, passive surveillance might not identify all myocarditis/myopericarditis cases after COVID-19 vaccination and it is possible that a mild/subclinical myocarditis might be much more prevalent in the population. This research project has three aims: first, provide novel insights regarding the incidence, patient characteristics and outcome of myocarditis. Second, provide a safety net by active surveillance for myocarditis, allowing early initiation of appropriate therapy. Third, provide reassurance to the public regarding myocarditis, as questions have been raised by critics of the pharmaceutical industry that Phase III studies performed by the pharmaceutical industry may have not appropriately captured adverse events.

This study is screening persons undergoing the COVID-19 mRNA booster vaccination of possible development of myocarditis. This approach in detecting myocarditis would help early initiation of the right treatment under close monitoring of the clinical course. Furthermore, this kind of study might also help understand the development of myocarditis and possibly the reasons for sex differences. Myocarditis suspicion is raised when patients present symptoms of acute chest discomfort, myalgia, fever/chills, abnormal ECG, increased concentrations of high-sensitivity cardiac troponin T (hs-cTnT), possibly supported by signs of cardiac inflammation in cMRI (myocardial oedema, myocardial/pericardial late gadolinium enhancement, pericardial effusion). Since the study is performed on health care professionals working in the University Hospital Basel, it is able to monitor more closely the possible side effects of the mRNA vaccination. Consecutive individuals that received a COVID-19 mRNA vaccine booster and undergo a systematic approach to detect myocarditis at the University Hospital Basel will be included.

ELIGIBILITY:
Inclusion Criteria:

* individuals working at the University Hospital Basel, Switzerland
* informed consent available
* 16-65 years old

Exclusion Criteria:

* Refusal to participate at the study
* Cardiac events or cardiac surgery within 30 days prior to study (as these could result in prolonged hs-cTnT elevations and interfere with the diagnosis of myocarditis

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive individuals that received a COVID-19 mRNA vaccine booster and undergo a systematic approach to detect myocarditis at the University Hospital Basel will be included. The project population includes mainly healthcare workers, aged between 16-65.
Sampling Method: Probability Sample
Enrollment: 835 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Incidence of myocarditis after mRNA COVID-19 mRNA booster vaccine | Assessment at day 3 (48- 96h) post-vaccination
  The primary endpoint is centrally adjudicated myocarditis after mRNA COVID-19 mRNA vaccine by a cardiologist according to current European Society of Cardiology (ESC) guidelines.

SECONDARY OUTCOMES:
Number of participants developing symptoms after the COVID-19 booster | Assessment at day 3 (48- 96h) post-vaccination
  Number of participants developing symptoms after the COVID-19 booster
Number of participants with MRI abnormalities after COVID-19 booster | Assessment at day 4 post-vaccination
  Number of participants with MRI abnormalities after COVID-19 booster
Composite of major adverse cardiac events | 1-month follow-up post-vaccination
  MACE is defined as a composite of acute heart failure (requiring admission to a hospital or intra-hospital transfer to the intensive care unit), cardiac death, life-threatening arrhythmia (cardiac arrest, sustained ventricular tachycardia, AV-block III), signs of left bundle branch block (LBBB) within 1 month after mRNA COVID-19 vaccination.
Need for hospitalization | At day 4 post-vaccination
  Need for hospitalization
Need for medical treatment | At day 4 post-vaccination
  Medical treatment could include, nonsteroidal anti-inflammatory medication (NSAIDs), use of immunomodulatory therapy such as colchicine (in cases with presumed pericardial inflammation) and intravenous globulins or corticosteroids, paracetamol, or morphine.
hs-cTnT/I concentrations on day 4 | At day 4 post-vaccination
  hs-cTnT/I concentrations on day 4
Total sum of costs (CHF) | 1-month follow-up post-vaccination
  Total sum of costs from involved study personnel, blood sampling, material used and further diagnostic work-up and treatment to estimate the financial value related to future screening of individuals receiving mRNA vaccines.
T cell reactivity | Assessment at day 4 post-vaccination
  T cell reactivity (against the SARS-CoV2 Spike, protein, myosin) in EDTA blood

CONTACTS AND LOCATIONS:
Overall Officials: Christian Müller, Prof. Dr. med., Principal Investigator — University Hospital Basel, Department of Cardiology
Locations (1):
- University Hospital Basel, Department of Cardiology, Basel, Switzerland